CLINICAL TRIAL: NCT04688671
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Study to Evaluate the Efficacy and Safety of ETX 018810 in Subjects With Diabetic Peripheral Neuropathic Pain
Brief Title: Efficacy and Safety of ETX-018810 for the Treatment of Diabetic Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eliem Therapeutics (UK) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETX-018810-202
Record Dates: First submitted 2020-12-25; First posted 2020-12-30 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Diabetic Peripheral Neuropathic Pain; Diabetic Peripheral Neuropathy

STUDY DESIGN:
Intervention Model Description: Placebo-Controlled, Parallel-Group
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ETX-018810 (Experimental): 1000 mg BID for 4 weeks
  Interventions: Drug: ETX-018810
- Placebo (Placebo Comparator): matching placebo BID for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ETX-018810 — Study Drug
  Arms: ETX-018810
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group Study to Evaluate the Efficacy and Safety of ETX 018810 in Subjects with Diabetic Peripheral Neuropathic Pain.

DETAILED DESCRIPTION:
ETX-018810 is a new chemical entity that is under development as a non-opioid treatment for chronic pain syndromes. ETX-018810 is a prodrug of palmitoylethanolamide (PEA), an endogenous bioactive lipid that has shown efficacy in a broad range of nonclinical inflammatory and neuropathic pain models and in clinical trials in chronic pain indications, including diabetic peripheral neuropathic pain (DPNP).

ELIGIBILITY:
Inclusion Criteria:

* The subject is ≥18 and ≤75 years of age at the time of signing ICF.
* The subject has a diagnosis of type 1 or 2 diabetes mellitus.
* The subject has diabetic neuropathy of a symmetrical nature in the lower extremities for ≥6 months to ≤10 years
* The subject reports at least moderate pain intensity
* The subject's onset of neuropathic pain is at least 3 months before the screening visit.
* The subject has used a stable regimen of antidiabetic agents for at least 1 month before the baseline visit or has achieved adequate glycemic control through diet and exercise.
* The subject has clinical laboratory values within normal limits or abnormal values that the investigator deems not clinically significant.
* Sexually active male subjects with female partners of childbearing potential and sexually active female subjects of childbearing potential must agree to practice effective contraception or to remain abstinent during the study and for 4 weeks after the last dose of investigational product
* The subject is capable of giving signed informed consent and agrees to provide authorization for use and release of health records.

Exclusion Criteria:

* The subject has pain that cannot be clearly differentiated from or that could interfere with the assessment of DPNP.
* The subject has neurologic and/or circulatory disorders that are unrelated to diabetic neuropathy
* The subject has a history of hypoglycemia that disturbed consciousness or ketoacidosis that required hospitalization within the 3 months before screening.
* The subject has clinically significant and/or unstable renal, hepatic, hematologic, immunologic, inflammatory/rheumatologic, respiratory, or cardiovascular disease that would compromise participation in the study in the judgment of the investigator.
* The subject has any neurological disease that could interfere with participation in the study (eg, Huntington's disease, Parkinson's disease, Alzheimer's disease, multiple sclerosis, seizures, epilepsy, stroke).
* The subject has an amputation of a lower extremity. Toe amputation is allowed.
* The subject has clinically significant abnormal electrocardiogram (ECG) findings at screening or baseline.
* The subject is likely to require major surgery during the study.
* The subject is pregnant or lactating.
* The subject is unwilling or unable to discontinue current medications for neuropathic pain, including topical agents.
* The subject is unable to refrain from using nonsteroidal anti-inflammatory drugs (NSAIDs); antiepileptic drugs, steroids, cannabinoids, or major opioids, muscle relaxants, tramadol, or tapentadol throughout the study.
* The subject has used prohibited nonpharmacologic therapies, including acupuncture, transcutaneous electrical nerve stimulation, etc, within 30 days before baseline/Day 1 or anticipates use of such therapies during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Delta Clinical Research, Mobile, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - Neuro-Pain Medical Cneter, Fresno, California
  - Encompass Clinical Research, Spring Valley, California
  - Diabetes Research Center, Tustin, California
  - Chase Medical Research LLC, Hamden, Connecticut
  - Charter Research, Lady Lake, Florida
  - Cordova Research Institute, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Better Health Clinical Reseach, Newnan, Georgia
  - Medisphere Medical Research Center, Evansville, Indiana
  - StudyMetrix Research LLC, City of Saint Peters, Missouri
  - Alliance for Multispeciality Research LLC, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - IMA Clinical Research, New York, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - FutureSearch Trials of Neurology, Austin, Texas
  - Alpine Research Organization, Clinton, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ETX-018810 | Placebo
Started | 83 | 84
Completed | 75 | 80
Not Completed | 8 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETX-018810 | Placebo | Total
Number analyzed (Participants) | 83 | 84 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 55 | 112
  >=65 years | 26 | 29 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (9.33) | 60.3 (9.87) | 60.4 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 34 | 59
  Male | 58 | 50 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 10 | 13 | 23
  White | 70 | 65 | 135
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 83 | 84 | 167
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.9 (4.33) | 30.9 (4.77) | 31.4 (4.57)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 4 in the Weekly Average of the Daily Pain Score as Derived From the Subject's Responses on the Pain Intensity Numerical Rating Scale (PI-NRS)
Description: Change from baseline in the weekly average of the daily pain score as derived from the subject's responses on the Pain Intensity Numerical Rating Scale (PI-NRS) a 10 point scale from 0 being the least (No Pain) to 10 being the most (Worst Possible Pain).
Time Frame: baseline to Week 4
Population: The modified ITT population included all randomized subjects who received at least one dose of study treatment and had at least four post-baseline PI-NRS measurements; 78 and 81 subjects for the ETX-018810 and Placebo groups, respectively. All subjects in this population were included in the statistical analysis comparing the groups. However, the descriptive summary for Week 4 only included those subjects who had measurements at Baseline and Week 4 (74 and 78 subjects, respectively).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 74 | 78
score on a scale | -1.79 (2.099) | -1.91 (1.781)
Statistical Analysis 1: Comparison: ETX-018810 vs Placebo; Test type: Superiority; p = 0.5605, Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 90% CI 2-sided [-0.32 to 0.68], Standard Error of Mean 0.302

2. Secondary Outcome: Number of Subjects With a ≥50% Reduction From Baseline to Weeks 1, 2, 3, and 4 in the Weekly Average of the Daily Pain Score
Description: Change in the weekly average of the daily pain score as derived from the subject's responses on the Pain Intensity Numerical Rating Scale (PI-NRS) a 10 point scale from 0 being the least (No Pain) to 10 being the most (Worst Possible Pain).
Time Frame: Baseline to Weeks 1, 2, 3 and 4
Population: The modified ITT population included all randomized subjects who received at least one dose of study treatment and had at least four post-baseline PI-NRS measurements; 78 and 81 subjects for the ETX-018810 and Placebo groups, respectively. Not all subjects had assessments at each week.
Measure: Count of Participants; unit: Participants
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 78 | 81
Participants
  Week 1: number analyzed (Participants) | 78 | 80
  Week 1 | 5 | 1
  Week 2: number analyzed (Participants) | 76 | 79
  Week 2 | 15 | 7
  Week 3: number analyzed (Participants) | 75 | 80
  Week 3 | 16 | 18
  Week 4: number analyzed (Participants) | 74 | 78
  Week 4 | 16 | 25

3. Secondary Outcome: Number of Subjects With a ≥30% Reduction From Baseline to Weeks 1, 2, 3, and 4 in the Weekly Average of the Daily Pain Score
Description: as for outcome 2
Time Frame: Baseline to Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 78 | 81
Participants
  Week 1: number analyzed (Participants) | 78 | 80
  Week 1 | 11 | 9
  Week 2: number analyzed (Participants) | 76 | 79
  Week 2 | 21 | 26
  Week 3: number analyzed (Participants) | 75 | 80
  Week 3 | 25 | 38
  Week 4: number analyzed (Participants) | 74 | 78
  Week 4 | 26 | 42

4. Secondary Outcome: Change in the Weekly Average of the Daily Pain Score From Baseline to Weeks 1, 2, and 3
Description: as for outcome 2
Time Frame: Baseline to Weeks 1, 2 and 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 78 | 81
score on a scale
  Week 1: number analyzed (Participants) | 78 | 80
  Week 1 | -0.67 (1.294) | -0.51 (1.009)
  Week 2: number analyzed (Participants) | 76 | 79
  Week 2 | -1.39 (1.879) | -1.16 (1.420)
  Week 3: number analyzed (Participants) | 75 | 80
  Week 3 | -1.60 (1.945) | -1.56 (1.682)

5. Secondary Outcome: Number of Subjects With a CGI-C Response (Defined as "Much Improved" or "Very Much Improved") at Week 4
Description: The Clinical Global Impression - Change (CGI-C) is a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to the baseline state at the beginning of the intervention. The rater selects one response based on the following question, "Compared to your patient's condition at the beginning of treatment, how much has your patient changed?" Scores are as follows: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Week 4
Population: The ITT population included all randomized subjects who received at least one dose of study treatment; 83 and 84 subjects for the ETX-018810 and Placebo groups, respectively. Not all subjects had a CGI-C assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 81 | 83
Participants | 26 | 34

6. Secondary Outcome: Number of Subjects With a PGI-C Response (Defined as "Much Improved" or "Very Much Improved") at Week 4.
Description: The Patient Global Impression - Change (PGI-C) is the patient-reported counterpoint to the CGI C (Guy, 1976). The qualitative assessment of meaningful change is determined by the patient in response to the question, "Compared to your condition at the beginning of treatment, how much has your condition changed?" Scores are as follows: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; and 7 = very much worse.
Time Frame: Week 4
Population: The ITT population included all randomized subjects who received at least one dose of study treatment; 83 and 84 subjects for the ETX-018810 and Placebo groups, respectively. Not all subjects in the population had a PGI-C assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 81 | 83
Participants | 27 | 37

7. Secondary Outcome: Change in the Weekly Average of the Daily Sleep Score on the DSIS From Baseline to Weeks 1, 2, 3, and 4
Description: The Daily Sleep Interference Scale (DSIS) is an 11-point response scale that quantifies sleep interference due to pain. It is a single-item measure that is completed once daily, upon awakening, to accurately capture variability in sleep interference due to pain on a daily basis, thus minimizing recall bias. Patients are asked to select the number that best describes how much their pain has interfered with their sleep during the last 24 hours on a scale from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep).
Time Frame: Baseline to Weeks 1, 2, 3 and 4
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 78 | 81
score on a scale
  Week 1: number analyzed (Participants) | 78 | 80
  Week 1 | -0.86 (1.554) | -0.67 (1.133)
  Week 2: number analyzed (Participants) | 76 | 79
  Week 2 | -1.36 (1.967) | -1.34 (1.480)
  Week 3: number analyzed (Participants) | 75 | 80
  Week 3 | -1.65 (2.087) | -1.73 (1.720)
  Week 4: number analyzed (Participants) | 73 | 78
  Week 4 | -1.70 (2.144) | -1.95 (1.900)

8. Secondary Outcome: Change in the BPI - Interference Scale From Baseline to Week 4
Description: The BPI Interference scale measures how much pain has interfered with seven daily activities scored on a scale from 0 (does not interfere) to 10 (completely interferes). It is scored as the mean of the seven interference items.
Time Frame: Baseline to Week 4
Population: The ITT population included all randomized subjects who received at least one dose of study treatment; 83 and 84 subjects for the ETX-018810 and Placebo groups, respectively. Not all subjects had a BPI assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 81 | 83
score on a scale | -1.60 (2.142) | -1.78 (2.202)

9. Secondary Outcome: Change in the BPI-Pain Scale From Baseline to Week 4
Description: The BPI pain scale is a composite of 4 items assessing pain severity (worst, least, average, and right now). Subjects rate their pain in last 24 hours on a scale from 0 (no pain) to 10 (pain as bad as you can imagine). It is scored as the mean of the four pain items.
Time Frame: Baseline to Week 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 81 | 83
score on a scale | -1.39 (1.833) | -1.78 (1.809)

10. Secondary Outcome: Change in the Daily Amount of Acetaminophen Use From Baseline to Week 4
Description: The daily amount of acetaminophen (rescue medication) that was used (mg per day).
Time Frame: Baseline to week 4
Population: The modified ITT population included all randomized subjects who received at least one dose of study treatment and had at least four post-baseline PI-NRS measurements; 78 and 81 subjects for the ETX-018810 and Placebo groups, respectively.
Measure: Median (Inter-Quartile Range); unit: mg per day
Arm/Group | ETX-018810 | Placebo
Number analyzed (Participants) | 78 | 81
mg per day | 0 [-105.9 to 0] | 0 [-92.9 to 0]

ADVERSE EVENTS:
Time Frame: 9 weeks (up to 4 week screening period, 4 week treatment period, & 1 week follow up period)
Arm/Group | ETX-018810 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/84
Serious Adverse Events (participants affected / at risk) | 1/83 | 0/84
Other Adverse Events (participants affected / at risk) | 22/83 | 11/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETX-018810 (N=83) | Placebo (N=84)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETX-018810 (N=83) | Placebo (N=84)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis astroviral (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the PI will provide the sponsor with a copy of any proposed communication at least 90 days in advance of the proposed submission or presentation date. Within this 90 day period, the sponsor will review the communication to determine whether it contains any sponsor Confidential Information, or whether the sponsor desires to file patent applications on subject matter contained therein, and to ensure the accuracy of the information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT04688671/Prot_SAP_001.pdf